CLINICAL TRIAL: NCT01947361
Title: Heterogeneity in Association of Heart Rate and Initial Presentation of Cardiovascular Diseases Using Linked Electronic Health Records
Brief Title: Heart Rate and Initial Presentation of Cardiovascular Diseases (Caliber)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Harry Hemingway, Professor, University College, London
Other Study IDs: 12_153R_IP10; RP-PG-0407-10314 (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Abdominal Aortic Aneurysm; Coronary Heart Disease NOS; Unheralded Coronary Death; Intracerebral Haemorrhage; Heart Failure; Ischemic Stroke; Myocardial Infarction; Stroke; Peripheral Arterial Disease; Stable Angina Pectoris; Subarachnoid Haemorrhage; Transient Ischemic Attack; Unstable Angina; Cardiac Arrest, Sudden Cardiac Death
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Cerebral Hemorrhage; Heart Failure; Ischemic Stroke; Myocardial Infarction; Stroke; Peripheral Arterial Disease; Angina, Stable; Subarachnoid Hemorrhage; Ischemic Attack, Transient; Angina, Unstable; Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study of heterogeneity in associations between heart rate and the initial presentation of 12 cardiovascular diseases.

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* One year prior to study entry (up-to-standard follow-up, CPRD quality research standard).
* > 30 years old
* have at least a recorded heart rate measurement during the study period

Exclusion Criteria:

- Evidence of prior atherosclerotic or cardiac disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1,96 million patients registered in Clinical Practice Research Datalink (CPRD) practices
Sampling Method: Non-Probability Sample
Enrollment: 1961286 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Risk of atherosclerotic disease in patients with high or low heart rate | Participants were followed until the first Coronary disease event (an expected average of 5 years)
  Hazard ratios will be also presenting associations between heart rate and initial presentation of different cardiovascular diseases. These associations will be also measured between different levels of heart rate and CVDs stratified by:
  * by sex
  * gender
  * a range of risk factors (such as physical activity, smoking status, drinking status, etc.)

SECONDARY OUTCOMES:
Incidence proportions and life time risk for Cardiovascular diseases | Participants were followed until the first Coronary disease event (an expected average of 5 years)
  Subhazard Ratios and Cumulative Incidence estimation of the risk of 12 different cardiovascular diseases adjusted for the 4 different levels of heart rate (<60, 60-74, 75-89, >90), age and sex in a lifetime period

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

REFERENCES:
- [Derived] Archangelidi O, Pujades-Rodriguez M, Timmis A, Jouven X, Denaxas S, Hemingway H. Clinically recorded heart rate and incidence of 12 coronary, cardiac, cerebrovascular and peripheral arterial diseases in 233,970 men and women: A linked electronic health record study. Eur J Prev Cardiol. 2018 Sep;25(14):1485-1495. doi: 10.1177/2047487318785228. Epub 2018 Jul 2. PMID 29966429
- See also: Related Info — http://www.caliberresearch.org/